CLINICAL TRIAL: NCT00447772
Title: Multicentre Open Study on the Efficacy and Safety of Botulinum Toxin A (500 Units Dysport®) in the Treatment of Heterogeneous Forms of Cervical Dystonia
Brief Title: Study to Assess the Efficacy and Safety of Dysport® in Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-94-52120-098; 2004-002086-20 (EudraCT Number)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Cervical Dystonia
Keywords: Dysport, Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Active Drug: Botulinum type A toxin (Dysport®) 500 Units / 2.5 ml injected in muscles involved in cervical dystonia
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The aim is to demonstrate equivalent efficacy and safety in the treatment of the two most frequent forms of cervical dystonia (predominantly rotational torticollis and predominantly laterocollis) with the standard initial dose of 500 units Dysport®. The patients will be assigned to one of the two basic types of cervical dystonia, either predominantly rotational torticollis or predominantly laterocollis on the basis of clinical examination. This will determine which therapy is to be administered, using the clearly defined, structured injection protocols.

ELIGIBILITY:
Inclusion Criteria:

* De novo patients with cervical dystonia
* Outpatient
* Patients to be of age 18 years or older
* Written informed consent to participate in the study

Exclusion Criteria:

* Pre-treatment of cervical dystonia with botulinum toxin
* Pre-treatment with botulinum toxin for any indication other than cervical dystonia within the past 12 months
* Pure retro- or antecollis
* Neurological or other diseases which may affect head and neck motor function or neuromuscular transmission, e.g. polyneuropathy with pareses, myasthenia, myopathy, motor neurone diseases, Bekhterev's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2004-10; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (105):
- Austria (5):
  - Krankenhaus der Barmherzigen Brüder, Graz
  - NÖ LKH Grimmenstein-Hochegg, Grimmenstein
  - Univ.-Klinik für Neurologie, Innsbruck
  - Konventhospital der Barmherzigen Brüder, Linz
  - O.Ö. Landes-Nervenklinik Wagner-Jauregg, Linz
- Germany (100):
  - Neurolog. Klinik des RWTH Aachen, Aachen
  - Praxis für Anästhesiologie, Ahaus
  - Praxis für Neurologie und Psychiatrie, Apolda
  - Sächsisches Krankenhaus, Arnsdorf
  - Praxis für Neurologie, Aschaffenburg
  - Klinikum für Rehabilitation, Bad Oeynhausen
  - Praxis für Neurologie, Bad Reichenhall
  - Krankenhaus Hohe Warte, Bayreuth
  - Neurologische Rehabilitationsklinik, Beelitz
  - NRZ Neurologisches Rehabilitationszentrum Leipzig, Bennewitz
  - Praxis für Neurologie, Berlin
  - Neurologisches Facharztzentrum am St.-Gertrauden-KH, Berlin
  - Universitätsklinikum Charité, Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Charité, Campus Virchow-Klinikum, Berlin
  - Gemeinschaftspraxis für Neurologie, Berlin
  - Krankenhaus Henningsdorf, Berlin
  - SALUS Fachkrankenhaus Bernburg, Bernburg
  - Neurologische Klinik GILEAD im Evang. KH Bielefeld EVKB, Bielefeld
  - Praxis für Neurologie, Bochum
  - Berufsg. Kliniken Bergmannsheil, Bochum
  - St.-Josef-Hospital, Bochum
  - Medizinische Einrichtung Rhein. F.-Wilhelms-Universität Bonn, Bonn
  - Zentralkrankenhaus Bremen-Ost, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Koeln-Merheim, Cologne
  - Praxis für Neurologie, Dachau
  - Bezirksklinikum Mainkofen, Deggendorf
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Malteser Krankenhaus St. Anna, Duisburg
  - University Hospital, Neurology Clinic, Düsseldorf
  - Landesklinik Eberswalde, Eberswalde
  - HELIOS Klinikum Erfurt, Erfurt
  - Uniklinik Erlangen, Erlangen
  - Alfried-Krupp-Krankenhaus, Essen
  - Universitätsklinik Essen, Essen
  - Kreiskrankenhaus Freiberg, Freiberg
  - Zentrum für Neurologie, Giessen
  - Praxis für Neurologie, Giessen
  - Praxis für Neurologie und Psychiatrie, Giessen
  - Sächsisches Krankenhaus für Psychiatrie, Psychotherapie und Neurolgie, Großschweidnitz
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Klinikum Ambrock, Hagen
  - Katholisches Krankenhaus Hagen, Hagen
  - Städt. Krankenhaus Martha-Maria, Halle
  - Gemeinschaftspraxis für Neurologie, Hamburg
  - Praxis für Neurologie, Hamburg
  - Neurologische Uniklinik, Hanover
  - Praxis für Neurologie, Hanover
  - Universitätskliniken des Saarlandes, Homburg
  - Gemeinschaftspraxis für Neurologie/Psychiatrie, Ilmenau
  - Praxis für Neurologie, Itzehoe
  - Uniklinik Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Universitätsklinikum Kiel, Kiel
  - Kath. Klinikum/Brüderkrankenhaus, Koblenz
  - Neurologische Praxis, Landshut
  - Universitätsklinikum Leipzig, Leipzig
  - Gemeinschaftspraxis für Neurologie/Psychiatrie, Leipzig
  - Gemeinschaftspraxis für Neurologie, Leipzig
  - Klinikum Lippe-Lemgo GmbH, Lemgo
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Universitätsklinikum, Lübeck
  - Gemeinschaftspraxis für Neurologie/Psychiatrie, Lüneburg
  - Universitätsklinikum, Magdeburg
  - Universitätsklinikum, Mainz
  - Klinikum Mannheim, Mannheim
  - Praxis für Neurologie, Mannheim
  - Klinikum Minden, Minden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Neurologisches Krankenhaus München, München
  - Klinikum rechts der Isar, München
  - Universitätsklinikum Münster, Münster
  - Praxis für Neurologie und Nervenheilkunde, Neubrandenburg
  - Klinikum Nürnberg-Süd, Nuremberg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Praxis für Neurologie und Psychiatrie, Ostfildern
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - St.-Josefs-Krankenhaus, Potsdam
  - Klinikum Ernst von Bergmann, Potsdam
  - Zentrum für Psychiatrie Weissenau, Ravensburg
  - Knappschafts-Krankenhaus, Recklinghausen
  - Universitätsklinikum, Rostock
  - Evang.-Freichkirchl. Krankenhaus, Rüdersdorf
  - Praxis für Neurologie, Schorndorf
  - Klinikum Uckermark GmbH, Schwedt
  - HELIOS Kliniken Schwerin, Schwerin
  - Asklepios Kliniken Schildautal, Seesen
  - EMSA, Singen
  - Landesfachkrankenhaus für Psychatrie und Neurologie, Stadtroda
  - Praxis für Neurologie, Stralsund
  - Neurologische Praxis, Straubing
  - Landesklinik Teupitz, Teupitz
  - Zentrum für Neurologie und Hertie-Institut für Klinische Hirnforschung, Tübingen
  - Klinikum Weiden, Weiden
  - Stiftung Deutsche Klinik für Diagnostik, Wiesbaden
  - Gemeinschaftspraxis für Neurologie, Wolfenbüttel
  - Klinikum Wuppertal, Wuppertal
  - Medizinisches Studienzentrum, Würzburg
  - Universitätsklinikum Würzburg, Würzburg
  - Paracelsus Klinik, Zwickau

REFERENCES:
- [Result] Hefter H, Benecke R, Erbguth F, Jost W, Reichel G, Wissel J. An open-label cohort study of the improvement of quality of life and pain in de novo cervical dystonia patients after injections with 500 U botulinum toxin A (Dysport). BMJ Open. 2013 Apr 18;3(4):e001853. doi: 10.1136/bmjopen-2012-001853. Print 2013. PMID 23604344
- [Result] Hefter H, Kupsch A, Mungersdorf M, Paus S, Stenner A, Jost W; Dysport Cervical Dystonia Study Group. A botulinum toxin A treatment algorithm for de novo management of torticollis and laterocollis. BMJ Open. 2011 Jan 1;1(2):e000196. doi: 10.1136/bmjopen-2011-000196. PMID 22021883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled (signed informed consent) 28 Oct 2004, last patient completed 4 April 2008. 516 patients were recruited to this prospective, open, multicentre study at 77 study centres in Germany and 4 study centres in Austria.
Pre-assignment Details: To be eligible patients had to have 2 of the most frequent forms of cervical dystonia (CD): rotatory torticollis or laterocollis.
Groups:
- Dysport® 500 U - Total Study Population: Patients with heterogeneous forms of CD were given a single intramuscular (i.m.) injection of 500 units (U) Dysport® at the first study visit (Week 0). The single injection of 500 U Dysport® was diluted in 2.5 millilitres (ml) 0.9% sodium chloride (= 200 units/ml). Patients were treated according to one of 12 possible basic patterns of injection protocol to allow individual treatment of the muscles affected as well as providing an algorithm for the individual first treatments.
  The patients visited the study centres at Week 4 and Week 12 post-dose for safety and efficacy assessments.
Period: Overall Study
Arm/Group | Dysport® 500 U - Total Study Population
Started | 516
Completed | 489
Not Completed | 27
Not completed — Lack of Efficacy | 3
Not completed — Insufficient compliance | 6
Not completed — Discontinuation of drug therapy | 1
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 1
Not completed — Unable to attend all study visits | 2
Not completed — Adverse Event | 1
Not completed — Patient relocated | 1
Not completed — Incomplete documentation at visit 1 | 1
Not completed — Chemotherapy for lung cancer | 1
Not completed — Premature re-injection required | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Population which included all patients who received the study medication and for who any safety data were recorded. All 516 patients who were enrolled received study medication. However, for one patient no safety data were available for analysis.
Groups:
- Dysport® 500 U - Total Study Population: Patients with heterogeneous forms of CD were given a single i.m. injection of 500 U Dysport® at the first study visit (Week 0). The single injection of 500 U Dysport® was diluted in 2.5 ml 0.9% sodium chloride (= 200 units/ml). Patients were treated according to one of 12 possible basic patterns of injection protocol to allow individual treatment of the muscles affected as well as providing an algorithm for the individual first treatments.
  The patients visited the study centres at Week 4 and Week 12 post-dose for safety and efficacy assessments.
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 353
  Male | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Score of the Tsui Rating Scale (Patient in Sitting Position) at the First On-treatment Visit (Week 4 or Week 12)
Description: The Tsui rating scale measures severity and duration of head deviation, shoulder elevation and head tremor. This instrument is based on 4 subscores:
  * Subscore A: amplitude of rotation, deflection (tilt) and ante- / retrocollis (range: 0-9 points)
  * Subscore B: duration of movement (values 1 or 2)
  * Subscore C: severity and duration of shoulder elevation (range: 0-3 points)
  * Subscore D: severity and duration of tremor (range: 0-4 points).
  The total score was calculated as follows: total score = subscores (A x B) + C + D. The total score ranges between 0 and 25 points. A high total score represents severe CD.
  The mean change in the total score of the Tsui rating scale (patient in the sitting position) between baseline (Week 0 visit) and the first on-treatment visit (Week 4 or Week 12 visit) is presented.
Time Frame: Baseline to Week 4 or Week 12 (up to 12 weeks)
Population: The Intention to Treat (ITT) Population included all patients in the safety population with a baseline visit (Week 0) and a post-baseline (Week 4 or Week 12) assessment of the Tsui rating scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rotatory Torticollis: Patients with rotatory torticollis type of CD who received a single i.m. injection of 500 U Dysport®.
- Laterocollis: Patients with laterocollis type of CD who received a single i.m. injection of 500 U Dysport®.
Arm/Group | Rotatory Torticollis | Laterocollis | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 396 | 107 | 503
units on a scale | -3.8 (3.3) | -4.0 (2.6) | -3.8 (3.1)
Statistical Analysis 1: Comparison: Rotatory Torticollis vs Laterocollis; An analysis of covariance (ANCOVA) model included the baseline total Tsui score (patient in sitting position) as covariate and the main type of CD as between-group factor (due to non-significance the interaction between baseline total Tsui score and the main type of CD was removed from the model); Test type: Superiority or Other; p = 0.2552, ANCOVA; Mean difference = -0.322, 95% CI 2-sided [-0.877 to 0.233] — The comparative analysis is based on adjusted means data

2. Secondary Outcome: Change in the Total Score of the Tsui Rating Scale (Patient in Sitting Position) Between Visit 1 (Week 0) and Visit 3 (Week 12)
Description: The Tsui rating scale measures severity and duration of head deviation, shoulder elevation and head tremor. This instrument is based on 4 subscores:
  * Subscore A: amplitude of rotation, deflection (tilt) and ante- / retrocollis (range: 0-9 points)
  * Subscore B: duration of movement (values 1 or 2)
  * Subscore C: severity and duration of shoulder elevation (range: 0-3 points)
  * Subscore D: severity and duration of tremor (range: 0-4 points).
  The total score was calculated as follows: total score = subscores (A x B) + C + D. The total score ranges between 0 and 25 points. A high total score represents severe CD.
  The mean change in the total score of the Tsui rating scale (patient in the sitting position) between baseline (Week 0 visit) and the Week 12 visit is presented.
Time Frame: Baseline to Week 12
Population: The ITT Population included all patients in the safety population with a baseline visit (Week 0) and a post-baseline (Week 4 or Week 12) assessment of the Tsui rating scale. Only patients with data available for the Week 12 visit are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotatory Torticollis | Laterocollis | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 386 | 104 | 490
units on a scale | -2.3 (3.4) | -2.4 (2.5) | -2.3 (3.2)

3. Secondary Outcome: Change in the Total Score of the Tsui Rating Scale (Patient Walking) Between Baseline (Week 0) and Visit 2 (Week 4) and Visit 3 (Week 12)
Description: The Tsui rating scale measures severity and duration of head deviation, shoulder elevation and head tremor. This instrument is based on 4 subscores:
  * Subscore A: amplitude of rotation, deflection (tilt) and ante- / retrocollis (range: 0-9 points)
  * Subscore B: duration of movement (values 1 or 2)
  * Subscore C: severity and duration of shoulder elevation (range: 0-3 points)
  * Subscore D: severity and duration of tremor (range: 0-4 points).
  The total score was calculated as follows: total score = subscores (A x B) + C + D.
  The total score ranges between 0 and 25 points. A high total score represents severe CD.
  The mean changes in the total score of the Tsui rating scale (patient walking) between baseline (Week 0 visit) and the Week 4 and Week 12 visits are presented.
Time Frame: Baseline to Week 4 and Week 12
Population: The ITT Population included all patients in the safety population with a baseline visit (Week 0) and a post-baseline (Week 4 or Week 12) assessment of the Tsui rating scale. Only patients with data available for each indicated timepoint are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotatory Torticollis | Laterocollis | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 396 | 107 | 503
units on a scale
  Change to Week 4 in total Tsui score: number analyzed (Participants) | 294 | 77 | 371
  Change to Week 4 in total Tsui score | -3.8 (3.2) | -4.3 (2.9) | -3.9 (3.2)
  Change to Week 12 in total Tsui score: number analyzed (Participants) | 285 | 79 | 364
  Change to Week 12 in total Tsui score | -2.3 (3.6) | -2.3 (3.1) | -2.3 (3.5)

4. Secondary Outcome: Change in the 4 Subscores of the Tsui Rating Scale (Patient in the Sitting Position) Between Visit 1 (Week 0) and Visit 2 (Week 4) and Visit 3 (Week 12)
Description: The Tsui rating scale measures severity and duration of head deviation, shoulder elevation and head tremor. This instrument is based on 4 subscores:
  * Subscore A: amplitude of rotation, deflection (tilt) and ante- / retrocollis (range: 0-9 points)
  * Subscore B: duration of movement (values 1 or 2)
  * Subscore C: severity and duration of shoulder elevation (range: 0-3 points)
  * Subscore D: severity and duration of tremor (range: 0-4 points).
  A higher score for each subscale represents severe CD symptoms. The total score was calculated as follows: total score = subscores (A x B) + C + D. The total score ranges between 0 and 25 points. A high total score represents severe CD.
  The mean changes in the subscores A to D of the Tsui rating scale (patient in the sitting position) between baseline (Week 0 visit) and the Week 4 and Week 12 visits are presented.
Time Frame: Baseline to Week 4 and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotatory Torticollis | Laterocollis | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 396 | 107 | 503
units on a scale
  Change to Week 4 in Tsui rating scale subscore A: number analyzed (Participants) | 394 | 106 | 500
  Change to Week 4 in Tsui rating scale subscore A | -1.3 (1.3) | -1.5 (1.2) | -1.4 (1.3)
  Change to Week 4 in Tsui rating scale subscore B: number analyzed (Participants) | 394 | 106 | 500
  Change to Week 4 in Tsui rating scale subscore B | -0.4 (0.6) | -0.3 (0.5) | -0.3 (0.6)
  Chang to Week 4 in Tsui rating scale subscore C: number analyzed (Participants) | 394 | 106 | 500
  Chang to Week 4 in Tsui rating scale subscore C | -0.4 (0.8) | -0.6 (0.8) | -0.4 (0.8)
  Change to Week 4 in Tsui rating scale subscore D: number analyzed (Participants) | 394 | 106 | 500
  Change to Week 4 in Tsui rating scale subscore D | -0.6 (1.0) | -0.5 (1.0) | -0.6 (1.0)
  Change to Week 12 in Tsui rating scale subscore A: number analyzed (Participants) | 386 | 104 | 490
  Change to Week 12 in Tsui rating scale subscore A | -0.8 (1.3) | -0.9 (1.2) | -0.8 (1.3)
  Change to Week 12 in Tsui rating scale subscore B: number analyzed (Participants) | 386 | 104 | 490
  Change to Week 12 in Tsui rating scale subscore B | -0.2 (0.5) | -0.1 (0.4) | -0.2 (0.5)
  Change to Week 12 in Tsui rating scale subscore C: number analyzed (Participants) | 386 | 104 | 490
  Change to Week 12 in Tsui rating scale subscore C | -0.2 (0.8) | -0.3 (0.7) | -0.2 (0.8)
  Change to Week 12 in Tsui rating scale subscore D: number analyzed (Participants) | 386 | 104 | 490
  Change to Week 12 in Tsui rating scale subscore D | -0.4 (0.9) | -0.3 (0.9) | -0.4 (0.9)

5. Secondary Outcome: Change in the Craniocervical Dystonia Questionnaire (CDQ-24) Total Score and Subscores Between Visit 1 (Week 0) and Visit 2 (Week 4) and Visit 3 (Week 12)
Description: The CDQ-24 is a disease-specific quality of life (QoL) instrument and was assessed at Visits 1 to 3. It consists of 24 items investigating problems in daily living skills related to CD.
  This instrument is based on 5 subscales: Stigma, Emotional well-being, Pain, Activities of daily living (ADL), Social/family life to which a number of the 24 items are assigned. There are five possible answers to each item representing increasing severity of impairment (scores 0 to 4). The total scores ranged from 0 to 96 (best to worst QoL). In order to obtain scores of the individual subscales, the total score of each subscale (sum of the individual item scores) was transformed linearly to a 0 to 100 scale (best to worst QoL).
  The mean changes in the CDQ-24 total score between baseline (Week 0 visit) and the Week 4 and Week 12 visits are presented.
Time Frame: Baseline to Week 4 and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 503
units on a scale
  Change to Week 4 in CDQ-24 total score: number analyzed (Participants) | 484
  Change to Week 4 in CDQ-24 total score | -11.1 (16.1)
  Change to Week 4 in CDQ-24 Stigma subscale: number analyzed (Participants) | 485
  Change to Week 4 in CDQ-24 Stigma subscale | -16.8 (24.0)
  Change to Week 4 in CDQ-24 Emotional subscale: number analyzed (Participants) | 485
  Change to Week 4 in CDQ-24 Emotional subscale | -10.3 (19.9)
  Change to Week 4 in CDQ-24 Pain subscale: number analyzed (Participants) | 491
  Change to Week 4 in CDQ-24 Pain subscale | -11.5 (27.8)
  Change to Week 4 in CDQ-24 ADL subscale: number analyzed (Participants) | 483
  Change to Week 4 in CDQ-24 ADL subscale | -11.1 (19.6)
  Change to Week 4 in CDQ-24 Social subscale: number analyzed (Participants) | 481
  Change to Week 4 in CDQ-24 Social subscale | -5.6 (17.9)
  Change to Week 12 in CDQ-24 total score: number analyzed (Participants) | 474
  Change to Week 12 in CDQ-24 total score | -11.8 (14.6)
  Change to Week 12 in CDQ-24 Stigma subscale: number analyzed (Participants) | 476
  Change to Week 12 in CDQ-24 Stigma subscale | -16.4 (22.5)
  Change to Week 12 in CDQ-24 Emotional subscale: number analyzed (Participants) | 476
  Change to Week 12 in CDQ-24 Emotional subscale | -11.1 (18.7)
  Change to Week 12 in CDQ-24 Pain subscale: number analyzed (Participants) | 484
  Change to Week 12 in CDQ-24 Pain subscale | -13.2 (25.5)
  Change to Week 12 in CDQ-24 ADL subscale: number analyzed (Participants) | 474
  Change to Week 12 in CDQ-24 ADL subscale | -12.5 (18.6)
  Change to Week 12 in CDQ-24 Social life subscale: number analyzed (Participants) | 469
  Change to Week 12 in CDQ-24 Social life subscale | -6.7 (17.8)

6. Secondary Outcome: Changes in the Items of the Patient Diary Based on Day-to-day Function and Activities, Pain and Duration of Pain Between Visit 1 (Week 0) and Visit 2 (Week 4) and Visit 3 (Week 12)
Description: The weekly recorded patient diary consists of the three items: Day-to-Day Capacities and Activities, Pain and Duration of Pain. Each item was rated by the patient on an 11-point scale ranging from 0 = no problems at all to 10 = most severe problems (the actual wording is adapted to each item in question).
  The mean changes between the baseline (Week 0 visit) and the Week 4 and Week 12 visits are presented.
Time Frame: Baseline to Week 4 and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 503
units on a scale
  Change to Week 4 in Day-to-day functions: number analyzed (Participants) | 454
  Change to Week 4 in Day-to-day functions | -1.1 (3.0)
  Change to Week 4 in Pain: number analyzed (Participants) | 452
  Change to Week 4 in Pain | -0.8 (2.7)
  Change to Week 4 in Duration of pain: number analyzed (Participants) | 451
  Change to Week 4 in Duration of pain | -1.2 (2.9)
  Change to Week 12 in Day-to-day functions: number analyzed (Participants) | 384
  Change to Week 12 in Day-to-day functions | -1.1 (2.6)
  Change to Week 12 in Pain: number analyzed (Participants) | 383
  Change to Week 12 in Pain | -0.9 (2.5)
  Change to Week 12 in Duration of pain: number analyzed (Participants) | 382
  Change to Week 12 in Duration of pain | -1.3 (2.7)

7. Secondary Outcome: Categorical Changes in the Items of the Patient Diary Based on Day-to-day Function and Activities, Pain and Duration of Pain Between Visit 1 (Week 0) and Visit 2 (Week 4) and Visit 3 (Week 12)
Description: The weekly recorded patient diary consists of the three items: Day-to-Day Capacities and Activities, Pain and Duration of Pain. Each item was rated by the patient on an 11-point scale ranging from 0 = no problems at all to 10 = most severe problems (the actual wording is adapted to each item in question).
  The following categorical changes between the baseline (Week 0 visit) and the Week 4 and Week 12 visits are presented: Improvement, No change and Deterioration.
Time Frame: Baseline to Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 503
percentage of patients
  Improvement in Day-to-day functions to Week 4: number analyzed (Participants) | 454
  Improvement in Day-to-day functions to Week 4 | 59.9
  No change in Day-to-day functions to Week 4: number analyzed (Participants) | 454
  No change in Day-to-day functions to Week 4 | 19.6
  Deterioration in Day-to-day functions to Week 4: number analyzed (Participants) | 454
  Deterioration in Day-to-day functions to Week 4 | 20.5
  Improvement in Pain to Week 4: number analyzed (Participants) | 452
  Improvement in Pain to Week 4 | 50.2
  No change in Pain to Week 4: number analyzed (Participants) | 452
  No change in Pain to Week 4 | 23.0
  Deterioration in Pain to Week 4: number analyzed (Participants) | 452
  Deterioration in Pain to Week 4 | 26.8
  Improvement in Duration in pain to Week 4: number analyzed (Participants) | 451
  Improvement in Duration in pain to Week 4 | 52.3
  No change in Duration of pain to Week 4: number analyzed (Participants) | 451
  No change in Duration of pain to Week 4 | 24.6
  Deterioration in Duration of pain to Week 4: number analyzed (Participants) | 451
  Deterioration in Duration of pain to Week 4 | 23.1
  Improvement in Day-to-day functions to Week 12: number analyzed (Participants) | 384
  Improvement in Day-to-day functions to Week 12 | 55.2
  No change in Day-to-day functions to Week 12: number analyzed (Participants) | 384
  No change in Day-to-day functions to Week 12 | 22.9
  Deterioration in Day-to-day functions to Week 12: number analyzed (Participants) | 384
  Deterioration in Day-to-day functions to Week 12 | 21.9
  Improvement in Pain to Week 12: number analyzed (Participants) | 383
  Improvement in Pain to Week 12 | 48.3
  No change in Pain to Week 12: number analyzed (Participants) | 383
  No change in Pain to Week 12 | 25.1
  Deterioration in Pain to Week 12: number analyzed (Participants) | 383
  Deterioration in Pain to Week 12 | 26.6
  Improvement in Duration of pain to Week 12: number analyzed (Participants) | 382
  Improvement in Duration of pain to Week 12 | 55.2
  No change in Duration of pain to Week 12: number analyzed (Participants) | 382
  No change in Duration of pain to Week 12 | 24.3
  Deterioration in Duration of pain to Week 12: number analyzed (Participants) | 382
  Deterioration in Duration of pain to Week 12 | 20.4

8. Secondary Outcome: Number of Patients Without Pain and/or With a Reduction in Pain Based on a Global Assessment of Pain by the Investigator and by the Patient at Visit 2 (Week 4) and Visit 3 (Week 12)
Description: Global pain was assessed at Visit 2 (Week 4) and Visit 3 (Week 12); investigators and patients assessed change in global pain according to the following response categories:
  1. = no pain (anymore)
  2. = less pain
  3. = no change
  4. = more pain
  The numbers of patients falling under each of these categories as assessed by the investigator and patient at Weeks 4 and 12 are presented.
Time Frame: Week 4 visit and Week 12 visit
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 503
Participants
  No pain at Week 4 (Investigator assessment): number analyzed (Participants) | 500
  No pain at Week 4 (Investigator assessment) | 131
  Less pain at Week 4 (Investigator assessment): number analyzed (Participants) | 500
  Less pain at Week 4 (Investigator assessment) | 205
  No change at Week 4 (Investigator assessment): number analyzed (Participants) | 500
  No change at Week 4 (Investigator assessment) | 94
  More pain at Week 4 (Investigator assessment): number analyzed (Participants) | 500
  More pain at Week 4 (Investigator assessment) | 70
  No pain at Week 12 (Investigator assessment): number analyzed (Participants) | 489
  No pain at Week 12 (Investigator assessment) | 142
  Less pain at Week 12 (Investigator assessment): number analyzed (Participants) | 489
  Less pain at Week 12 (Investigator assessment) | 227
  No change at Week 12 (Investigator assessment): number analyzed (Participants) | 489
  No change at Week 12 (Investigator assessment) | 87
  More pain at Week 12 (Investigator assessment): number analyzed (Participants) | 489
  More pain at Week 12 (Investigator assessment) | 33
  No pain at Week 4 (Patient assessment): number analyzed (Participants) | 500
  No pain at Week 4 (Patient assessment) | 128
  Less pain at Week 4 (Patient assessment): number analyzed (Participants) | 500
  Less pain at Week 4 (Patient assessment) | 202
  No change at Week 4 (Patient assessment): number analyzed (Participants) | 500
  No change at Week 4 (Patient assessment) | 82
  More pain at Week 4 (Patient assessment): number analyzed (Participants) | 500
  More pain at Week 4 (Patient assessment) | 88
  No pain at Week 12 (Patient assessment): number analyzed (Participants) | 490
  No pain at Week 12 (Patient assessment) | 132
  Less pain at Week 12 (Patient assessment): number analyzed (Participants) | 490
  Less pain at Week 12 (Patient assessment) | 231
  No change at Week 12 (Patient assessment): number analyzed (Participants) | 490
  No change at Week 12 (Patient assessment) | 83
  More pain at Week 12 (Patient assessment): number analyzed (Participants) | 490
  More pain at Week 12 (Patient assessment) | 44

9. Secondary Outcome: Global Assessment of Efficacy by the Investigator and by the Patient at Visit 2 (Week 4) and Visit 3 (Week 12)
Description: At Visit 2 (Week 4) and Visit 3 (Week 12) investigators and patients assessed global efficacy of injection of 500 U Dysport® according to the following response categories:
  1. = very good
  2. = good
  3. = moderate
  4. = insufficient
  The numbers of patients falling under each of these categories as assessed by the investigator and patient at Weeks 4 and 12 are presented.
Time Frame: Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dysport® 500 U - Total Study Population
Number analyzed (Participants) | 503
Participants
  Week 4 (Investigator assessment): Very good: number analyzed (Participants) | 500
  Week 4 (Investigator assessment): Very good | 129
  Week 4 (Investigator assessment): Good: number analyzed (Participants) | 500
  Week 4 (Investigator assessment): Good | 221
  Week 4 (Investigator assessment): Moderate: number analyzed (Participants) | 500
  Week 4 (Investigator assessment): Moderate | 109
  Week 4 (Investigator assessment): Insufficient: number analyzed (Participants) | 500
  Week 4 (Investigator assessment): Insufficient | 41
  Week 12 (Investigator assessment): Very good: number analyzed (Participants) | 489
  Week 12 (Investigator assessment): Very good | 134
  Week 12 (Investigator assessment): Good: number analyzed (Participants) | 489
  Week 12 (Investigator assessment): Good | 218
  Week 12 (Investigator assessment): Moderate: number analyzed (Participants) | 489
  Week 12 (Investigator assessment): Moderate | 102
  Week 12 (Investigator assessment): Insufficient: number analyzed (Participants) | 489
  Week 12 (Investigator assessment): Insufficient | 35
  Week 4 (Patient assessment): Very good: number analyzed (Participants) | 500
  Week 4 (Patient assessment): Very good | 97
  Week 4 (Patient assessment): Good: number analyzed (Participants) | 500
  Week 4 (Patient assessment): Good | 207
  Week 4 (Patient assessment): Moderate: number analyzed (Participants) | 500
  Week 4 (Patient assessment): Moderate | 113
  Week 4 (Patient assessment): Insufficient: number analyzed (Participants) | 500
  Week 4 (Patient assessment): Insufficient | 83
  Week 12 (Patient assessment): Very good: number analyzed (Participants) | 490
  Week 12 (Patient assessment): Very good | 113
  Week 12 (Patient assessment): Good: number analyzed (Participants) | 490
  Week 12 (Patient assessment): Good | 205
  Week 12 (Patient assessment): Moderate: number analyzed (Participants) | 490
  Week 12 (Patient assessment): Moderate | 100
  Week 12 (Patient assessment): Insufficient: number analyzed (Participants) | 490
  Week 12 (Patient assessment): Insufficient | 72

ADVERSE EVENTS:
Time Frame: From Visit 1 (Week 0) to Visit 3 (Week 12) for each patient.
Description: All adverse events are reported as treatment emergent adverse events. The Safety Population includes all patients who received the study medication and for whom any safety data were recorded.
Arm/Group | Dysport® 500 U - Total Study Population
All-Cause Mortality (participants affected / at risk) | 0/515
Serious Adverse Events (participants affected / at risk) | 11/515
Other Adverse Events (participants affected / at risk) | 206/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 500 U - Total Study Population (N=515)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 500 U - Total Study Population (N=515)
Circulatory collapse (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Limb operation (Surgical and medical procedures) | 1 (1)
Asthenia (General disorders) | 3 (3)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Injection site pain (General disorders) | 7 (7)
Injection site paraesthesia (General disorders) | 1 (1)
Local swelling (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Sensation of foreign body (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Initial insomnia (Psychiatric disorders) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Blood pressure orthostatic abnormal (Investigations) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 4 (4)
Cervical root pain (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 12 (13)
Dysarthria (Nervous system disorders) | 4 (4)
Head discomfort (Nervous system disorders) | 2 (2)
Head titubation (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 17 (21)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Mastication disorder (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4)
Paralysis (Nervous system disorders) | 1 (1)
Paresis (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2)
Tongue paralysis (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Blepharitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eyelid ptosis (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Keratoconjunctivitis sicca (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 51 (51)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 70 (70)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (12)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 34 (35)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 1 (1)
Eye infection viral (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 2 (2)
Laryngitis (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 19 (20)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less